CLINICAL TRIAL: NCT05685368
Title: The Healing Power of Acceptance: Evaluating the Efficacy of Acceptance and Commitment Therapy (ACT) in Combating the Effects of Race-Related Stress Among Black Adolescents
Brief Title: Acceptance and Commitment Therapy (ACT) for Combating the Effects of Race-Related Stress Among Black Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Xzania Lee, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-23-00089
Record Dates: First submitted 2023-01-05; First posted 2023-01-17 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Race-related Stress; Depression, Anxiety; Quality of Life; Stress Reaction
Keywords: Black; African American; Adolescents; Acceptance and Commitment Therapy; race-related stress; racial trauma; coping
MeSH Terms: conditions — Depression; Anxiety Disorders; Fractures, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Acceptance Commitment Therapy (Experimental): This study will use a 10-session ACT protocol to support Black adolescents and young adults in coping with race related stress.
  Interventions: Behavioral: ACT for Race Related Stress

INTERVENTIONS:
Behavioral: ACT for Race Related Stress — This intervention will be guided by: Payne, J. S. (2022). Out of the Fire: Healing Black Trauma Caused by Systemic Racism Using Acceptance and commitment Therapy New Harbinger Publications, Inc.

SUMMARY:
The current study seeks to build on previous research that demonstrates the efficacy of Acceptance and Commitment Therapy in combating stigma by investigating the feasibility and acceptability of a protocol to support Black adolescents and young adults in coping with race related stress. The study will consist of a small, purposeful, non-randomized sample (N = 30) of clients enrolled into a 10-session Acceptance and Commitment Therapy group. The group will be offered as part of regular clinical care at the Division of Adolescent and Young Adult Medicine. Three consecutive groups will be run with approximately 8-10 participants in each group over the next year.

ELIGIBILITY:
Inclusion Criteria:

* Identify as Black/African American
* English-speaking

Exclusion Criteria:

* Prisoners or youth in detention centers will be excluded.
* Not capable of participating meaningfully in the assent/consent process.
* Being at significant risk for suicide and self-injury
* Currently experiencing psychosis
* Having severe health concerns that will impact study participation or attendance

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Total Score on Index of Race-Related Stress (IRRS)-Brief Version | 12 weeks
  Higher scores on this measure indicate greater race-related stress. The minimum score on this measure is 0 and the maximum is 88.

SECONDARY OUTCOMES:
Total Scores on Acceptance and Action Questionnaire-2 | 12 weeks
  Higher scores on this measure indicate greater psychological flexibility. The minimum score on this measure is 7 and the maximum is 49.
Total Scores on Multidimensional Inventory of Black Identity-Teen (MIBI-t) | 12 weeks
  Higher scores on this measure indicate stronger racial identity. The minimum score on this measure is 21 and the maximum is 105.
Total Score on Patient Health Questionaire-9 | 12 weeks
  Higher scores indicate greater depression. The minimum score on this measure is 0 and the maximum is 27.
Total Score on General Anxiety Disorder-7 | 12 weeks
  Higher scores indicate greater anxiety. The minimum score on this measure is 0 and the maximum is 21.

CONTACTS AND LOCATIONS:
Overall Officials: Xzania Lee, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No